CLINICAL TRIAL: NCT06453681
Title: Dexmedetomidine As an Adjuvant to Bupivacaine in Bilateral Pectoral Nerve Blocks for Postoperative Pain Control After Cardiac Surgeries: a Randomized Controlled Trial
Brief Title: Dexmedetomidine As an Adjuvant to Bupivacaine in Bilateral PECs for Pain Control After Cardiac Surgeries
Acronym: PECs
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Assisstent professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MD-75-2024
Record Dates: First submitted 2024-05-27; First posted 2024-06-12 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain
Keywords: PECs; dexameditomedine
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bupivacain (Active Comparator): patients receive bilateral Pecs block with bupivacin 0.25%,
  Interventions: Other: bilateral PECS
- dexameditomedine bupivacain (Active Comparator): patients received bilateral Pecs block with bupivacin 0.25% plus dexmedetomidine 0.5 μg/Kg as adjuvant.
  Interventions: Other: bilateral PECS; Drug: Dexmedetomidine

INTERVENTIONS:
Other: bilateral PECS — ectoralis nerve (Pecs) block, which is novel, less invasive regional analgesic technique.
  Other Names: PECTORAL NERVE BLOCK
Drug: Dexmedetomidine — Dexmedetomidine is a potent α2 agonist. In our practice, dexmedetomidine is administered as an additive to regional anesthesia to improve the duration and quality of analgesia
  Other Names: precedex
  Arms: dexameditomedine bupivacain

SUMMARY:
the study aims to test the quality of analgesia provided by dexmedetomidine as an adjuvant to bupivacaine bilateral PECs block in patients scheduled for cardiothoracic surgeries with median sternotomy incision.

DETAILED DESCRIPTION:
Background: Good postoperative analgesia in cardiac surgical patients helps in early recovery and ambulation. An alternative to parenteral, paravertebral, and thoracic epidural analgesia can be pectoralis nerve (Pecs) block, which is a novel, less invasive regional analgesic technique.

The study aims to test the quality of analgesia provided by dexmedetomidine as an adjuvant to bupivacaine bilateral PECs block in patients scheduled for cardiothoracic surgeries with median sternotomy incision.

sixty adult patients between the age groups of 25 and 65 years undergoing coronary artery bypass grafting or valve surgeries through midline sternotomy under general anesthesia were enrolled in the study. Patients were randomly allocated into two groups with 30 ineach group. Group 1 patients will receive bilateral Pecs block, whereas Group 2 patients will receive bilateral Pecs block with dexameditomedine postoperatively. Patients will be extubated once they fulfilled extubation criteria. Ventilator duration will be recorded. Patients will be interrogated for pain by visual analog scale (VAS) scoring at rest and cough. Inspiratory flow rate will be assessed using incentive spirometry.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients between the age groups of 25 and 65 years undergoing either coronary artery bypass grafting (CABG) or valve surgeries through midline sternotomy under general anesthesia

Exclusion Criteria:

* Skin erosions, hematomas or infection at the injection site.
* coagulopathy, ACT more than 150 seconds
* History of hypersensitivity to bupivacaine or Dexametomedine.
* The Patients who are unable to use the pain score.
* patients who will need prolonged post-operative ventilation or inotropic support.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
The duration of analgesia | up to 24 hour
  from block start time (time of LA injection) to block end time at which VAS score 4 or more)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kasralainy school of medicine, Cairo
  - Kasralaini Faculty of Medicine, Cairo

IPD SHARING:
Plan to Share IPD: No